CLINICAL TRIAL: NCT01665131
Title: The Use of Subcutaneous Implantable Cardiac Defibrillators (ICDs) Following Extraction of Conventional ICDs
Acronym: SUBTRACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Manav Sohal, Clinical Research Fellow, Guy's and St Thomas' NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUBTRACT 1
Record Dates: First submitted 2012-08-10; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Use of Subcutaneous ICDs Following Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subcutaneous ICD group (Experimental)
  Interventions: Device: Cameron Health S-ICD SQ-RX

INTERVENTIONS:
Device: Cameron Health S-ICD SQ-RX

SUMMARY:
Implantable cardiac defibrillators (ICDs) are devices that are put into patients at high risk of sudden cardiac death. They are used to treat life threatening heart rhythm disorders. They have conventionally consisted of a generator sitting under the skin of the chest and leads which pass from veins in the collar bone region to the heart. Problems with these devices can necessitate extraction, with the commonest reason being infection. If extraction is required for infection then re-implantation is usually deferred for approximately one week whilst antibiotics are given so that the risk of infection of the new device can be minimised. This has considerable implications for healthcare resources. A new ICD has been developed that is entirely subcutaneous with no intravenous element. It is already in clinical use and is positioned remote from conventional ICD sites. With no intravenous element there is very little risk of infection in the blood affecting the new device. It is therefore likely to be possible to re-implant these devices immediately after extracting a conventional system. The aim of this research is to assess the outcome in patients re-implanted with this device immediately after conventional ICD system extraction. This data will be compared compared to those who have conventional systems re-implanted after the necessary delay.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling conventional criteria for ICD extraction and who require implantation of a further ICD without a need for pacing.

Exclusion Criteria:

* Indication for anti-bradycardia pacing or cardiac resynchronisation therapy
* Life expectancy < 1 year
* Need for intravenous inotropes
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay

SECONDARY OUTCOMES:
Rate of ICD infection | 1 year
  To see what the infection rate of new implants is and to assess how this compares to published rates of infection when using the standard method.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Rinaldi, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust